CLINICAL TRIAL: NCT00908531
Title: Randomized Trial of Endocrine Therapy Against Locoregional Therapy First. A DBCG Trial in Postmenopausal Patients With Operable Hormone Receptor Positive Tumors Larger Than 2 cm.
Brief Title: Trial of Endocrine Against Locoregional Therapy First in Postmenopausal Women With Early Breast Cancer
Acronym: REAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitement
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Collaborators: The Danish Medical Research Council (Other); Danish Cancer Society (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Bent Ejlertsen, Professor, MD, PhD, Danish Breast Cancer Cooperative Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBCG 07-REAL
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Operable Breast Neoplasms
Keywords: Breast neoplasms; Randomised trial; Aromatase Inhibitors; Preoperative care; Age 60 or older; Hormone receptor positive tumor; Tumor lager than 2 cm; No distant metastasis
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postoperative letrozole (Active Comparator): Definitive surgery without preoperative AI treatment
  Interventions: Drug: letrozole (Femara)
- Preoperative letrozole (Experimental): Treatment with letrozole for 4 months before definitive surgery.
  Interventions: Drug: letrozole (Femara)

INTERVENTIONS:
Drug: letrozole (Femara) — tablet 2.5 mg daily
  Other Names: Femara

SUMMARY:
The hypothesis to be addressed in this randomized phase III trial is that 4 months of letrozole may be superior to surgery as primary therapy for early stage hormone receptor positive breast cancer in postmenopausal women, provided that these patients will receive definitive and radical surgery and adjuvant therapies as otherwise indicated at the completion of preoperative letrozole.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 60 years or older
* Measurable non-metastatic and non-inflammatory breast cancer
* Tumor of 2 cm or larger
* ER and/or PgR positive tumor
* Co-morbidity index 0 - 3, e.g., no other serious medical condition

Exclusion Criteria:

* Prior medical therapy for a malignant disease, including aromatase inhibitors
* Distant metastasis
* Need for chemotherapy
* Past or current history of other neoplasms (except for curative treated basal skin cancer or in situ carcinoma of the cervix uteri)
* Treatment with a non-approved drug within 30 days

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2009-05; Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
pCR | At four months
  Complete response rate
Clinical tumor response | At four months
  Ultrasound

SECONDARY OUTCOMES:
Overall survival | At ten years
  Death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Bent Ejlertsen, MD, PhD, Principal Investigator — DBCG
Locations (9):
- Denmark (9):
  - Dept. of Breast Surgery; Aalborg Sygehus, Aalborg
  - Dept. of Surgery; Århus Sygehus, Aarhus
  - Dept. of Breast Surgery; Rigshospitalet, Copenhagen
  - Dept. of Surgery; Sydvestjysk Sygehus Esbjerg, Esbjerg
  - Dept. of Breast Surgery; Herlev Hospital, Herlev
  - Dept. of Oncology; Odense University Hospital, Odense
  - Depart. of Breast Surgery, Ringsted Sygehus, Ringsted
  - Dept. of Breast Surgery; Vejle Sygehus, Vejle
  - Dept. of Breast Surgery; Regionshospitalet Viborg, Viborg

REFERENCES:
- [Background] Skriver SK, Laenkholm AV, Rasmussen BB, Handler J, Grundtmann B, Tvedskov TF, Christiansen P, Knoop AS, Jensen MB, Ejlertsen B. Neoadjuvant letrozole for postmenopausal estrogen receptor-positive, HER2-negative breast cancer patients, a study from the Danish Breast Cancer Cooperative Group (DBCG). Acta Oncol. 2018 Jan;57(1):31-37. doi: 10.1080/0284186X.2017.1401228. Epub 2017 Nov 23. PMID 29168427
- [Derived] Skriver SK, Jensen MB, Knoop AS, Ejlertsen B, Laenkholm AV. Tumour-infiltrating lymphocytes and response to neoadjuvant letrozole in patients with early oestrogen receptor-positive breast cancer: analysis from a nationwide phase II DBCG trial. Breast Cancer Res. 2020 May 14;22(1):46. doi: 10.1186/s13058-020-01285-8. PMID 32410705